CLINICAL TRIAL: NCT02981030
Title: Acceptability and Feasibility of a Simplified Medical Abortion Service Delivery in Western Ukraine: A Demonstration Study of 800 mcg Buccal Misoprostol Following 200 mg Mifepristone for Abortion up to 70 Days Gestation
Brief Title: Acceptability and Feasibility of a Simplified Medical Abortion Service Delivery in Western Ukraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Charitable Foundation Women Health & Family Planning (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1037
Record Dates: First submitted 2016-11-16; First posted 2016-12-02 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Abortion, Therapeutic
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Simplified medical abortion (Experimental): Women seeking medical abortion will be offered the option self-administering the medications, mifepristone and misoprostol at home.
  Interventions: Drug: Mifepristone; Drug: Misoprostol

INTERVENTIONS:
Drug: Mifepristone — Women seeking medical abortion will be offered the option to take mifepristone at home
Drug: Misoprostol — Women seeking medical abortion will be offered the option to take misoprostol at home. Misoprostol will be administered buccally.

SUMMARY:
The study will examine how a simplified outpatient medical abortion procedure using mifepristone and misoprostol, with the option to take mifepristone at a place of woman's choosing, works in Ukraine. The investigators intend to demonstrate the efficacy of oral administration of 200 mg mifepristone and buccal administration of 800 mcg misoprostol with gestations through 70 days, as well as the acceptability of this method.

ELIGIBILITY:
Inclusion Criteria:

* Have an intrauterine pregnancy consistent with gestational age less than 71 days;
* Be able to understand and willing to sign a consent form;
* Be eligible for medical abortion according to the clinician's assessment;
* Be able to return to the clinic and able to contact study staff or emergency medical services, if needed;
* Be willing to provide an address and/or telephone number for purposes of follow-up;
* Agree to comply with the study procedures and visit schedule.

Exclusion Criteria:

* Confirmed or suspected ectopic pregnancy or undiagnosed adnexal mass;
* Chronic renal failure;
* Concurrent long-term corticosteroid therapy;
* History of allergy to mifepristone, or misoprostol or another prostaglandin;
* History of hemorrhagic disorders or concurrent anticoagulant therapy;
* History of inherited porphyrias;
* Intrauterine device in place (must be removed before mifepristone is administered).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-11-23 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of successful abortion | 2 weeks after mifepristone administration

CONTACTS AND LOCATIONS:
Overall Officials: Ingrida Platais, MS, Principal Investigator — Gynuity Health Projects; Tamar Tsereteli, MD, MSc, PhD, Principal Investigator — Gynuity Health Projects; Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Galyna Maystruk, MD, Study Director — Charitable Foundation Women Health & Family Planning
Locations (2):
- Ukraine (2):
  - Lviv Municipal Women's Consultation No. 2, Lviv
  - Vinnitsa Regional Clinical Hospital, Vinnitsa

IPD SHARING:
Plan to Share IPD: No